CLINICAL TRIAL: NCT03159286
Title: Experimental Test of Facebook Social Drinking Norms on Adolescent Alcohol Use
Acronym: Network
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of North Texas Health Science Center (Other)
Responsible Party: Principal Investigator, Dana Litt, Affiliate Associate Professor, University of North Texas Health Science Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 50829
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Feedback, Psychological; Underage Alcohol Use; Risk-Taking
MeSH Terms: conditions — Underage Drinking; Risk-Taking

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know which intervention they are in during the course of the study. They will be debriefed at the end of the study and informed which condition they were a part of.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Abstainer (Experimental): Participants view social networking site profiles with alcohol content that references abstaining from alcohol use.
  Interventions: Behavioral: Abstainer
- Abstainer + User (Experimental): Participants view social networking site profiles with alcohol content that references both abstaining from alcohol use and using alcohol.
  Interventions: Behavioral: Abstainer + User
- Control (Experimental): Participants view social networking site profiles with no alcohol content.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Abstainer — Participants view social networking site profiles with alcohol content referencing abstaining from alcohol use.
  Arms: Abstainer
Behavioral: Abstainer + User — Participants view social networking site profiles with alcohol content referencing abstaining from alcohol use and using alcohol.
  Arms: Abstainer + User
Behavioral: Control — Participants view social networking site profiles with no alcohol content.
  Arms: Control

SUMMARY:
The proposed research will be the first study to focus on experimentally manipulating both injunctive and descriptive norms on social networking sites in order to elucidate the relationship between alcohol and abstainer displays on social networking sites and subsequent alcohol cognitions, use, and related negative consequences. Based on literature focusing on developmentally appropriate health models for adolescents, the Prototype Willingness Model (PWM) assumes that health-risk behaviors occur either when individuals have developed intentions to engage in a risk behavior (and these intentions vary as a function of attitudes and perceived injunctive norms) or through willingness to engage in risks (which varies as a function of perceived vulnerability to negative consequences, perceived descriptive norms , and prototypes). To fully understand the relationships between alcohol abstaining displays on social networking sites, we will examine 1) the role of descriptive and injunctive abstainer and user norms, when experimentally manipulated with SNS profiles, on willingness and intentions, subsequent alcohol use and related negative consequences among adolescents (age 1 5-20) 2) whether intentions and willingness mediate the relation between our experimental manipulation and subsequent alcohol use and negative consequences and whether 3) individual differences in social influence moderate the effect of the experimental manipulation on intentions, willingness, alcohol use, and negative consequences. We will test these aims by recruiting a community sample of adolescents (N = 300), living in the greater Seattle metropolitan area. Participants will complete a web-based baseline assessment and participate in an in-person experimental manipulation in which they are either assigned to see same-sex social networking site profiles of alcohol abstainers, abstainers +users, or a control condition where neither user or abstainer information will be provided. Immediately after the manipulation, participants will answer a series of questions about the profiles they just viewed and their alcohol-related cognitions. Participants will also complete a one-month in person follow up assessment to test for impacts on intentions, willingness, alcohol use, and related negative consequences. Additionally, individual differences in social influence will be examined as possible moderators o f the relationship between SNS-portrayed norms and our primary outcomes. This study is both significant and innovative in that it uses a theoretical perspective to experimentally test the impact of alcohol content, in particular abstainer norms, on Facebook on adolescent alcohol use and related cognitions. The results have the potential to inform preventative interventions while addressing NIH priorities.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 15 and 20 years old
* Must reside within Seattle area
* Must use alcohol at least once in the last 6 months
* Must have valid email address
* Must have active profile on social networking site (Facebook, Instagram and/or Snapchat)
* Regular access to the web or personal mobile phone
* Willing to come to office for the experimental manipulation and post-manipulation assessment.

Exclusion Criteria:

* The only exclusion criteria is not to not meet the above inclusion criteria

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 306 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Willingness and Intentions to Use Alcohol | Baseline, Post-Manipulation and 1-Month Follow-Up time points
  Assesses willingness to use alcohol and intentions to use alcohol at Baseline, Post-Manipulation, and 1-Month Follow-Up assessments.
Change in Self-Reported Alcohol Use | Baseline and 1-Month Follow-Up time points
  Assesses self-reported alcohol use (using the Daily Drinking Questionnaire and Quantity Frequency measures) at Baseline and 1-Month Follow-Up assessments.
Change in Alcohol-Related Negative Consequences | Baseline and 1-Month Follow-Up time points
  Assesses alcohol-related negative consequences (using the Young Adult Alcohol Consequences Questionnaire) at Baseline and 1-Month Follow Up.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for the Study of Health and Risk Behaviors, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
A select number of researchers will have access to unidentified participant data at the close of the study.